CLINICAL TRIAL: NCT03247426
Title: Comparison of Sleep Quality, Job Satisfaction, Quality of Life, Occupational Burnout Levels Among Individuals Who do or do Not do Exercise
Brief Title: Sleep Quality, Job Satisfaction, Quality of Life, Occupational Burnout Levels in Individuals
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: HACETTEPEUNIV
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Evaluation individuals with exercise: Individuals who work in sitting position and do regular exercises will be recruited.
  Interventions: Other: Evaluation individuals
- Evaluation individuals without exercise: Individuals who work in sitting position and do not perform regular exercises will be recruited.
  Interventions: Other: Evaluation individuals

INTERVENTIONS:
Other: Evaluation individuals — Sleep quality of the individuals, job satisfaction, quality of life, occupational burnout level will be evaluated.

SUMMARY:
The aim of this study is to compare sleep quality, job satisfaction, quality of life, occupational burnout levels among individuals who do or do not do exercise.

DETAILED DESCRIPTION:
Physical activity is very important in terms of healthy growth and development, protection from unwanted bad habits, socialization, protection from chronic diseases, and providing an active aging period. At the same time it increases the quality of life throughout life.Especially in individuals who work in sitting position, the risk of physical activity decrease due to intensive working hours, time constraint, social insufficiency is even more risk.Therefore, it is aimed to compare sleep quality, job satisfaction, quality of life, occupational burnout levels among individuals who do or do not do exercise.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals;

* Between the ages of 25-65 years,
* Those who are in the profession group working for at least 8 hours,
* who do the same job for at least 5 years,
* Individuals with no doctor-diagnosed skeletal system disease will be included.

Exclusion Criteria:

Individuals;

* Below the age of 25 years and above the age of 65 years,
* Individuals with doctor-diagnosed skeletal system disease will be excluded.

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy individuals who aged between 25-65 years, are in the profession group working for at least 8 hours, do the same job for at least 5 years, and having no doctor-diagnosed skeletal system disease will be included.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Sleep quality of the individuals | 15 days
  Pittsburgh Sleep Quality Index (PUKI) will be used to evaluate sleep quality.

SECONDARY OUTCOMES:
job satisfaction | 15 days
  Minnesota Job Satisfaction Scale (MIS) will be used to evaluate job satisfaction.
quality of life | 15 days
  World Health Organization Quality of Life Scale Short Form (WHOQOL-BREF) will be used to evaluate quality of life of the individuals.
occupational burnout level | 15 days
  Maslach Burnout Scale will be used to evaluate occupational burnout.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No